CLINICAL TRIAL: NCT01912677
Title: Oral Antihypertensive Regimens for Management of Hypertension in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Government Medical College, Nagpur (Industry); Daga Memorial Women's Hospital, Nagpur, India (Other); University of British Columbia (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4000
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Hypertension in Pregnancy; Preeclampsia
Keywords: hypertension in pregnancy; preeclampsia; anti-hypertension; labetalol; nifedipine; methyldopa
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Nifedipine; Labetalol; Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nifedipine (Active Comparator): Women will receive an initial dose of oral nifedipine 10mg. If blood pressure exceeds 155mmHg systolic OR 105 mmHg diastolic after 1h, an additional 10mg dose can be provided each hour for two additional doses (30 mg total).
  Interventions: Drug: Nifedipine
- Methyldopa (Experimental): Women will receive an initial dose of oral methyldopa 1000mg. No additional escalation in dose in the first 6 hours will be given.
  Interventions: Drug: Methyldopa
- Labetalol (Experimental): Women will receive an initial dose of oral labetalol 200mg. If blood pressure exceeds 155mmHg systolic OR 105 mmHg diastolic after 1h, an additional 200mg dose can be provided each hour for two additional doses (600 mg total).
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Nifedipine
  Arms: Nifedipine
Drug: Labetalol
  Arms: Labetalol
Drug: Methyldopa
  Arms: Methyldopa

SUMMARY:
This is a pragmatic, open-label, randomised control trial of three oral anti-hypertensive regimens for women with severe hypertension in pregnancy. Women presenting with severe hypertension in pregnancy in two hospitals in Nagpur, India will be randomised to one of three oral regimens: nifedipine, labetalol or methyldopa. This trial will compare the efficacy, safety and side effects of these three oral regimens for management of hypertension in pregnant women. The investigators hypothesize that nifedipine treatment of severe hypertensive parturient women is more effective than treatment with labetalol or methyldopa in controlling high blood pressure within six hours.

DETAILED DESCRIPTION:
This is a pragmatic, open-label, randomised control trial of three oral anti-hypertensive regimens for women with severe hypertension in pregnancy. Women presenting with severe hypertension in pregnancy in two hospitals in Nagpur, India will be randomised to one of three oral regimens: nifedipine, labetalol or methyldopa. This trial will compare the efficacy, safety and side effects of these three oral regimens for management of hypertension in pregnant women. The investigators hypothesize that nifedipine treatment of severe hypertensive parturient women is more effective than treatment with labetalol or methyldopa in controlling high blood pressure within six hours.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant gestational age >= 28 weeks
* Systolic blood pressure >=160 mm Hg OR a diastolic blood pressure of >=110 mm Hg measured twice more than 15 minutes apart
* Able to swallow pills
* >= 18 years

Exclusion Criteria:

* Indication for emergent cesarean or known fetal anomaly
* Anti-hypertensive therapy received in the past 12 hours
* History of eclampsia or other adverse CNS complication (e.g., stroke or PRES) in this pregnancy
* Actively wheezing at time of enrollment or history of asthma complications
* Known coronary artery disease or type I DM with microvascular complications or signs of heart failure or clinical dissection of the aorta

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 894 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Successful outcome | 6 hours
  Successful outcome will be considered blood pressure that reaches the target (defined as 120-150mmHg systolic and 70-100 mmHg mm Hg diastolic) at 6h without an adverse outcome.

SECONDARY OUTCOMES:
number of hourly BP's in severe range | one hour
  the number of hourly BP's in severe range

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Principal Investigator — Gynuity Health Projects
Locations (2):
- India (2):
  - Daga Women's Hospital, Nagpur, Maharashtra
  - Government Medical College, Nagpur, Maharashtra

REFERENCES:
- [Derived] Easterling T, Mundle S, Bracken H, Parvekar S, Mool S, Magee LA, von Dadelszen P, Shochet T, Winikoff B. Oral antihypertensive regimens (nifedipine retard, labetalol, and methyldopa) for management of severe hypertension in pregnancy: an open-label, randomised controlled trial. Lancet. 2019 Sep 21;394(10203):1011-1021. doi: 10.1016/S0140-6736(19)31282-6. Epub 2019 Aug 1. PMID 31378394